CLINICAL TRIAL: NCT04493203
Title: A Phase II Trial of Nivolumab Plus Axitinib in Patients With Anti-PD1 Refractory Advanced Melanoma
Brief Title: Nivolumab Plus Axitinib in Patients With Anti-PD1 Refractory Advanced Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yana Najjar (Other)
Collaborators: Pfizer (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Yana Najjar, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 20-101
Record Dates: First submitted 2020-07-22; First posted 2020-07-30 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Advanced Melanoma; Unresectable Melanoma
MeSH Terms: interventions — Nivolumab; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nivolumab plus Axitinib (Experimental): Nivolumab 480mg, IV, every 4 weeks, for up to two years.
  Axitinib 5mg, PO, BID, for up to two years.
  Interventions: Drug: Nivolumab; Drug: Axitinib

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is a human IgG4 monoclonal antibody that blocks PD-1. It is a type of Immunotherapy and works as a checkpoint inhibitor, blocking a signal that prevents activation of T cells from attacking the cancer.
  Other Names: Opdivo; AG013736
Drug: Axitinib — Axitinib (AG013736; trade name Inlyta) is a small molecule tyrosine kinase inhibitor.Its primary mechanism of action is thought to be vascular endothelial growth factor receptor 1-3, c-KIT and PDGFR inhibition, this, in turn, enables it to inhibit angiogenesis (the formation of new blood vessels by tumours)
  Other Names: INLYTA

SUMMARY:
This is Phase II trial of nivolumab plus axitinib for patients with unresectable stage III or IV melanoma who have progressed on prior anti-PD1 therapy with or without concomitant anti-CTLA4 therapy. Patients will receive treatment with nivolumab 480 mg intravenously every 4 weeks and axitinib 5 mg twice daily by mouth. Patients may continue both agents for up to two years if they do not experience disease progression or dose-limiting toxicities.

DETAILED DESCRIPTION:
This trial hypothesizes that decreasing hypoxia in the TME will re-sensitize melanoma tumors to anti-PD1 therapy. Axitinib has already been safely combined with anti-PD1 therapy and was overall well-tolerated. With nivolumab plus axitinib taken together, based on previously published work and data from our laboratories, it is hypothesized that axitinib can metabolically remodel the TME to render it more sensitive to ICB, specifically by reducing intra-tumoral hypoxia, increasing T cell infiltration, and increasing polyfunctional T cells. It will determined if treatment with nivolumab plus axitinib will prolong both progression-free and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Have unresectable (stage III) or advanced (stage IV) cutaneous or mucosal melanoma. Patients with uveal melanoma are not eligible.
* Progressed on prior anti-PD1 therapy with or without anti-CTLA4 therapy. Patients may have progressed in the adjuvant setting if treated within the last 6 months. Prior treatment with BRAF/MEK inhibitors permitted, however, not required. Progression must be radiographic, and progression of disease will be confirmed by a radiologist. Patients must have progressed during anti-PD-1 therapy, defined as unequivocal progression on or within 3 months of the last dose of anti-PD-1 therapy if treated in the metastatic setting, or within 6 months if treated in the adjuvant setting.
* Have measurable disease based on RECIST 1.1.
* Patients do not have to have biopsiable disease to be eligible. However, patients with biopsiable disease must undergo biopsy at study entry and at week 12.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Demonstrate adequate organ function, per protocol
* Patients with brain metastases are permitted if they are asymptomatic or previously treated with CNS directed therapy with stable CNS disease for at least 2 weeks. Stable is defined as asymptomatic or not progressing on imaging.
* Female patients of childbearing potential - negative pregnancy testing; use of birth control, surgically sterile or abstain from heterosexual activity during study and for 5 months after the last dose of study medication.
* Male subjects - agree to use an adequate contraception starting with the first dose of study therapy through 7 months after the last dose of study therapy; abstinence acceptable

Exclusion Criteria:

* Prior history of Grade 3 or 4 immune-related adverse events or immune-related adverse events requiring discontinuation of prior therapies.
* History of hypertensive crisis or hypertensive encephalopathy.
* Significant thrombotic (e.g. deep vein thrombosis or pulmonary embolism) or hemorrhagic event within 6 months prior to enrollment.
* History of prior immune-related adverse event due to an anti-PD1 or anti-CTLA4 that has not resolved to grade 1 on a steroid dose of prednisone 10 mg or less at the time of study entry (excluding vitiligo and endocrine toxicity).
* Patients with prior myocarditis or other immune-mediated cardiac adverse events, prior Guillain-Barre syndrome, encephalitis, meningitis, or transverse myelitis, prior Stevens-Johnson syndrome or toxic epidermal necrolysis are excluded regardless of grade.
* Poorly controlled hypertension defined as systolic blood pressure (SBP) > 160 and/or diastolic blood pressure (DBP) > 100 despite antihypertensives. If subject is above this goal, treatment with anti-hypertensives to achieve better blood pressure control is permitted. Ambulatory blood pressure assessment is permitted if there is concern for discrepant blood pressure readings while patients are in clinic.
* Has Class III or IV heart failure based on the New York Heart Association.
* Has had major surgery within 4 weeks of randomization. This does not include outpatient surgeries that do not require post-operative admission.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (greater than the equivalent of prednisone 10 mg daily, unless for prior endocrine toxicity) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment (premedication with steroids for contrast imaging studies is permitted).
* Has a known history of active TB (Bacillus Tuberculosis).
* Hypersensitivity to nivolumab or axitinib, or any of their excipients.
* Has had prior chemotherapy or targeted small molecule therapy within 1 week prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Has had radiation within 2 weeks of randomization.
* Has current use or anticipated need for treatment with drugs or foods that are known strong cytochrome P450 (CYP34A4/5) inhibitors including but not limited to atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, troleandomycin, voriconazole, and grapefruit or grapefruit juice. NOTE: The topical use of these medications, such as 2% ketoconazole cream is allowed.
* Has current use or anticipated need for treatment with drugs known to be strong CYP3A4/5 inducers, including but not limited to carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, and St. John's wort.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy, in situ cervical cancer, in situ colon cancer, or nonmetastatic prostate cancer not on systemic therapy.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 2 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has an active infection requiring systemic IV antibiotic therapy.
* Has had any of the following within the past 6 months
* Myocardial infarction or unstable angina
* Ventricular arrythmia
* Acute decompensated heart failure
* Cerebrovascular accident
* Hypertensive emergency requiring ICU admission
* Presence of a disorder that may impact absorption of axitinib, such as inability to take oral medication, requirement for IV alimentation, prior gastric resection, treatment for active peptic ulcer confirmed by endoscopy within the past 3 months, active GI bleed, malabsorption syndrome.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 5 months after the last dose of trial treatment for females and 7 months after the last dose of trial treatment for males.
* Has a known history of HIV (HIV 1/2 antibodies) if the CD4 count is less than 350 mm3 or serum HIV viral load is < 25,000 IU/mL.
* Has a known history of or is positive for hepatitis B (hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (hepatitis C virus [HCV] RNA [qualitative] is detected). Note: Without known history, testing only needs to be performed if there is clinical suspicion for Hepatitis B or C.
* Is currently incarcerated or otherwise detained.
* Has received a live vaccine within 30 days of planned start of study therapy. (intranasal iNinfluenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed)

Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.

Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2025-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yana Najjar, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nivolumab Plus Axitinib
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2903 (12.8924)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Percentage of patients who achieve Complete Response (CR) or Partial Response (PR) as best response by RECIST v1.1 criteria (with exact 95% CI). Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR) is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 31
percentage of patients | 10 [2 to 25.8]

2. Primary Outcome: Overall Response Rate (ORR) - Prior Ipilimumab / Nivolumab Treatment
Description: Percentage of patients (prior Ipilimumab/Nivolumab treatment) who achieve Complete Response (CR) or Partial Response (PR) as best response by RECIST v1.1 criteria (with exact 95% CI). Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR) is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients who were previously treated with Ipilimumab/Nivolumab and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 16
percentage of patients | 6.3 [0.2 to 30.2]

3. Primary Outcome: Overall Response Rate (ORR) - no Prior Ipilimumab / Nivolumab
Description: Percentage of patients (no prior Ipilimumab/Nivolumab treatment) who achieve Complete Response (CR) or Partial Response (PR) as best response by RECIST v1.1 criteria (with exact 95% CI). Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR) is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients who were not previously treated with Ipilimumab/Nivolumab and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 15
percentage of patients | 13.3 [1.7 to 40.5]

4. Primary Outcome: Overall Response Rate (ORR) - Prior Lines of Therapy <=3
Description: Percentage of patients (<=3 prior lines of therapy) who achieve Complete Response (CR) or Partial Response (PR) as best response by RECIST v1.1 criteria (with exact 95% CI). Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR) is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients who received <=3 prior lines of therapy and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 20
percentage of patients | 15 [3.2 to 37.9]

5. Primary Outcome: Overall Response Rate (ORR) - Prior Lines of Therapy >3
Description: Percentage of patients (>3 prior lines of therapy) who achieve Complete Response (CR) or Partial Response (PR) as best response by RECIST v1.1 criteria (with exact 95% CI). Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR) is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients who received >3 prior lines of therapy were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 11
percentage of patients | 0 [0 to 28.5]

6. Primary Outcome: Overall Response Rate (ORR) by iRECIST
Description: Percentage of patients with Complete Response (CR), Partial Response (PR), or Stable Disease (SD). Per iRECIST. (CR): disappearance of a target lesion. Any pathological lymph nodes (target or non-target) must have reduction in short axis to <10 mm. (PR): at least 30% decrease in sum of diameters of target lesions, with reference the baseline sum diameters. Can have had iUPD (one or more instances), but not iCPD, before iCR, iPR, or iSD
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 15
percentage of patients | 0 [0 to 21.8]

7. Primary Outcome: Overall Response Rate (ORR) - Primary IO Resistance
Description: Percentage of patients (with primary IO resistance) who achieve Complete Response (CR) or Partial Response (PR) as best response by RECIST v1.1 criteria (with exact 95% CI). Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR) is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 15
percentage of patients | 0 [0 to 21.8]

8. Primary Outcome: Overall Response Rate (ORR) - Secondary IO Resistance
Description: Percentage of patients (with secondary IO resistance) who achieve Complete Response (CR) or Partial Response (PR) as best response by RECIST v1.1 criteria (with exact 95% CI). Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR) is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 16
percentage of patients | 18.8 [4 to 45.6]

9. Primary Outcome: Overall Response Rate (ORR) - Acral Histology
Description: Percentage of patients (acral histology) who achieve Complete Response (CR) or Partial Response (PR) as best response by RECIST v1.1 criteria (with exact 95% CI). Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR) is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients with acral histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 7
percentage of patients | 14.3 [0.4 to 57.9]

10. Primary Outcome: Overall Response Rate (ORR) - Cutaneous Histology
Description: Percentage of patients (with cutaneous histology) who achieve Complete Response (CR) or Partial Response (PR) as best response by RECIST v1.1 criteria (with exact 95% CI). Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR) is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients with cutaneous histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 17
percentage of patients | 5.9 [0.1 to 28.7]

11. Primary Outcome: Overall Response Rate (ORR) - Mucosal Histology
Description: Percentage of patients (with mucosal histology) who achieve Complete Response (CR) or Partial Response (PR) as best response by RECIST v1.1 criteria (with exact 95% CI). Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR) is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients with mucosal histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 7
percentage of patients | 14.3 [0.4 to 57.9]

12. Primary Outcome: Disease Control Rate (DCR)
Description: Percentage of patients with Complete Response (CR), Partial Response (PR), or Stable Disease (SD). Per RECIST v1.1. (CR): the disappearance of a target lesion. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. (PR): at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. (SD): neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study.
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 31
percentage of patients | 45.2 [27.3 to 64.0]

13. Primary Outcome: Disease Control Rate (DCR) - no Prior Ipilimumab / Nivolumab Treatment
Description: as for outcome 12
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients who were not previously treated with Ipilimumab /Nivolumab and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 15
percentage of patients | 33.3 [11.8 to 61.6]

14. Primary Outcome: Disease Control Rate (DCR) - Prior Ipilimumab / Nivolumab Treatment
Description: as for outcome 12
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients who were previously treated with Ipilimumab /Nivolumab and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 16
percentage of patients | 56.3 [29.9 to 80.2]

15. Primary Outcome: Disease Control Rate (DCR) - Prior Lines of Therapy <=3
Description: Percentage of patients (<=3 prior lines of therapy) with Complete Response (CR), Partial Response (PR), or Stable Disease (SD). Per RECIST v1.1. (CR): the disappearance of a target lesion. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. (PR): at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. (SD): neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study.
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients who received<=3 prior lines of therapy and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 20
percentage of patients | 50 [27.2 to 72.8]

16. Primary Outcome: Disease Control Rate (DCR) - Prior Lines of Therapy >3
Description: Percentage of patients (>3 prior lines of therapy) with Complete Response (CR), Partial Response (PR), or Stable Disease (SD). Per RECIST v1.1. (CR): the disappearance of a target lesion. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. (PR): at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. (SD): neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study.
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients who received >3 prior lines of therapy and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 11
percentage of patients | 36.4 [10.9 to 69.2]

17. Primary Outcome: Disease Control Rate (DCR) by iRECIST
Description: Percentage of patients with Complete Response (CR), Partial Response (PR), or Stable Disease (SD). Per iRECIST. (CR): disappearance of a target lesion. Any pathological lymph nodes (target or non-target) must have reduction in short axis to <10 mm. (PR): at least 30% decrease in sum of diameters of target lesions, with reference the baseline sum diameters. (SD): neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, reference the smallest sum diameters while on study. Can have had iUPD (one or more instances), but not iCPD, before iCR, iPR, or iSD
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 15
percentage of patients | 40.0 [16.3 to 67.7]

18. Primary Outcome: Disease Control Rate (DCR) - Secondary IO Resistance
Description: Percentage of patients (with secondary IO resistance) with Complete Response (CR), Partial Response (PR), or Stable Disease (SD). Per RECIST v1.1. (CR): the disappearance of a target lesion. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. (PR): at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. (SD): neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study.
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients with secondary IO resistance who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 16
percentage of patients | 37.5 [15.2 to 64.6]

19. Primary Outcome: Disease Control Rate (DCR) - Primary IO Resistance
Description: Percentage of patients (with primary IO resistance) with Complete Response (CR), Partial Response (PR), or Stable Disease (SD). Per RECIST v1.1. (CR): the disappearance of a target lesion. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. (PR): at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. (SD): neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study.
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients with primary IO resistance who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 15
percentage of patients | 53.3 [26.6 to 78.7]

20. Primary Outcome: Disease Control Rate (DCR) - Acral Histology
Description: Percentage of patients (with acral histology) with Complete Response (CR), Partial Response (PR), or Stable Disease (SD). Per RECIST v1.1. (CR): the disappearance of a target lesion. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. (PR): at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. (SD): neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study.
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients with acral histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 7
percentage of patients | 71.4 [29.0 to 96.3]

21. Primary Outcome: Disease Control Rate (DCR) - Cutaneous Histology
Description: Percentage of patients (with cutaneous histology) with Complete Response (CR), Partial Response (PR), or Stable Disease (SD). Per RECIST v1.1. (CR): the disappearance of a target lesion. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. (PR): at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. (SD): neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study.
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients with cutaneous histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 17
percentage of patients | 35.3 [14.2 to 61.7]

22. Primary Outcome: Disease Control Rate (DCR) - Mucosal Histology
Description: Percentage of patients (with mucosal histology) with Complete Response (CR), Partial Response (PR), or Stable Disease (SD). Per RECIST v1.1. (CR): the disappearance of a target lesion. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. (PR): at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. (SD): neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study.
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients with mucosal histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 7
percentage of patients | 42.9 [9.9 to 81.6]

23. Primary Outcome: Best Response
Description: Percentage of patients with Complete Response (CR), Partial Response (PR), or Stable Disease (SD) or Progressive Disease (PD). Per RECIST v1.1. (CR): the disappearance of a target lesion. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. (PR): at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. (SD): neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study. (PD): at least a 20% increase in the sum of diameters of target lesions, taking as a reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (the appearance of one or more new lesions is also considered progression).
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients who were evaluable for radiologic response.
Measure: Number; unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 31
percentage of patients
  Partial Response | 10
  Stable Disease | 35
  Progressive Disease | 55

24. Primary Outcome: Best Response - no Prior Ipilimumab / Nivolumab
Description: as for outcome 23
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients who were not previously treated with Ipilimumab /Nivolumab and were evaluable for radiologic response.
Measure: Number; unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 15
percentage of patients
  Partial Response | 13.3
  Stable Disease | 20.0
  Progressive Disease | 66.7

25. Primary Outcome: Best Response - Prior Ipilimumab / Nivolumab Treatment
Description: as for outcome 23
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients who were previously treated with Ipilimumab/Nivolumab and were evaluable for radiologic response.
Measure: Number; unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 16
percentage of patients
  Partial Response | 6.3
  Stable Disease | 50.0
  Progressive Disease | 43.8

26. Primary Outcome: Best Response - Acral Histology
Description: Percentage of patients (with acral histology) with Complete Response (CR), Partial Response (PR), or Stable Disease (SD) or Progressive Disease (PD). Per RECIST v1.1. (CR): the disappearance of a target lesion. Any pathological lymph nodes (target or non-target) must have reduction in short axis to <10 mm. (PR): at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. (SD): neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study. (PD): at least a 20% increase in the sum of diameters of target lesions, taking as a reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (the appearance of one or more new lesions is also considered progression).
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients with acral histology who were evaluable for radiologic response.
Measure: Number; unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 7
percentage of patients
  Partial Response | 14.3
  Stable Disease | 57.1
  Progressive Disease | 28.6

27. Primary Outcome: Best Response - Cutaneous Histology
Description: Percentage of patients (with cutaneous histology) with Complete Response (CR), Partial Response (PR), or Stable Disease (SD) or Progressive Disease (PD). Per RECIST v1.1. (CR): the disappearance of a target lesion. Any pathological lymph nodes (target or non-target) with reduction in short axis to <10 mm. (PR): at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. (SD): neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study. (PD): at least a 20% increase in the sum of diameters of target lesions, taking as a reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (the appearance of one or more new lesions is also considered progression
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients with cutaneous histology who were evaluable for radiologic response.
Measure: Number; unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 17
percentage of patients
  Partial Response | 5.9
  Stable Disease | 29.4
  Progressive Disease | 64.7

28. Primary Outcome: Best Response - Mucosal Histology
Description: Percentage of patients (with mucosal histology) with Complete Response (CR), Partial Response (PR), or Stable Disease (SD) or Progressive Disease (PD). Per RECIST v1.1. (CR): the disappearance of a target lesion. Any pathological lymph nodes (target or non-target) with reduction in short axis to <10 mm. (PR): at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. (SD): neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study. (PD): at least a 20% increase in the sum of diameters of target lesions, taking as a reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (the appearance of one or more new lesions is also considered progression
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients with mucosal histology who were evaluable for radiologic response.
Measure: Number; unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 7
percentage of patients
  Partial Response | 14.3
  Stable Disease | 28.6
  Progressive Disease | 57.1

29. Primary Outcome: Best Response - Prior Lines of Therapy <=3
Description: Percentage of patients (<=3 prior lines of therapy) with Complete Response (CR), Partial Response (PR), or Stable Disease (SD) or Progressive Disease (PD). Per RECIST v1.1. (CR): the disappearance of a target lesion. Any pathological lymph nodes (target or non-target) must have reduction in short axis to <10 mm. (PR): at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. (SD): neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study. (PD): at least a 20% increase in the sum of diameters of target lesions, taking as a reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (the appearance of one or more new lesions is also considered progression).
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients who received <=3 prior lines of therapy and were evaluable for radiologic response.
Measure: Number; unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 20
percentage of patients
  Partial Response | 15.0
  Stable Disease | 35.0
  Progressive Disease | 50.0

30. Primary Outcome: Best Response - Prior Lines of Therapy >3
Description: Percentage of patients (>3 prior lines of therapy) with Complete Response (CR), Partial Response (PR), or Stable Disease (SD) or Progressive Disease (PD). Per RECIST v1.1. (CR): the disappearance of a target lesion. Any pathological lymph nodes (target or non-target) must have reduction in short axis to <10 mm. (PR): at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. (SD): neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study. (PD): at least a 20% increase in the sum of diameters of target lesions, taking as a reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (the appearance of one or more new lesions is also considered progression).
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients who received <=3 prior lines of therapy and were evaluable for radiologic response.
Measure: Number; unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 11
percentage of patients
  Partial Response | 0
  Stable Disease | 36.4
  Progressive Disease | 63.6

31. Primary Outcome: Best Response by iRECIST
Description: Percentage of patients with Complete Response (CR), Partial Response (PR), or Stable Disease (SD) or Progressive Disease (PD). Per iRECIST v1.1. (CR): the disappearance of a target lesion. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. (PR): at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. Can have had iUPD (one or more instances), but not iCPD, before iCR, iPR, or iSD
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients who were evaluable for radiologic response.
Measure: Number; unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 15
percentage of patients
  iCPD/iUPD | 60
  iSD | 40

32. Primary Outcome: Best Response - Primary IO Resistance
Description: Percentage of patients (w/ primary IO resistance) with Complete Response (CR), Partial Response (PR), or Stable Disease (SD) or Progressive Disease (PD). Per RECIST v1.1. (CR): the disappearance of a target lesion. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. (PR): at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. (SD): neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study. (PD): at least a 20% increase in the sum of diameters of target lesions, taking as a reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (the appearance of one or more new lesions is also considered progres
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients with primary IO resistance who were evaluable for radiologic response.
Measure: Number; unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 15
percentage of patients
  Partial Response | 0.0
  Stable Disease | 53.3
  Progressive Disease | 46.7

33. Primary Outcome: Best Response - Secondary IO Resistance
Description: Percentage of patients (w/ secondary IO resistance) with Complete Response (CR), Partial Response (PR), or Stable Disease (SD) or Progressive Disease (PD). Per RECIST v1.1. (CR): the disappearance of a target lesion. Any pathological lymph nodes (target or non-target) must have reduction in short axis to <10 mm. (PR): at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. (SD): neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study. (PD): at least a 20% increase in the sum of diameters of target lesions, taking as a reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (the appearance of one or more new lesions is also considered progres
Time Frame: Up to 12 weeks from baseline (after treatment)
Population: Treated patients with secondary IO resistance who were evaluable for radiologic response.
Measure: Number; unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 16
percentage of patients
  Partial Response | 18.8
  Stable Disease | 18.8
  Progressive Disease | 62.5

34. Secondary Outcome: Overall Survival (OS) - Overall Cohort
Description: The median number of months from the start of treatment that patients remain alive, until death from any cause.
Time Frame: Up to 45 months
Population: All enrolled patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 31
months | 10.0 [7.00 to 16.00]

35. Secondary Outcome: 6-month Overall Survival (OS)
Description: Percentage of patients alive from the start of treatment that patients remain alive, until death from any cause up to 6 months.
Time Frame: Up to12 months
Population: All enrolled patients.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 31
percentage of patients | 71 [52 to 84]

36. Secondary Outcome: 12-month Overall Survival (OS)
Description: Percentage of patients alive from the start of treatment that patients remain alive, until death from any cause up to 12 months.
Time Frame: Up to 12 months
Population: All enrolled patients.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 31
percentage of patients | 35 [19 to 52]

37. Secondary Outcome: 24-month Overall Survival (OS)
Description: Percentage of patients alive from the start of treatment that patients remain alive, until death from any cause up to 24 months.
Time Frame: Up to 24 months
Population: All enrolled patients.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 30
percentage of patients | 21 [9 to 37]

38. Secondary Outcome: Overall Survival (OS) - Prior Ipilimumab/Nivolumab Treatment
Description: The median number of months from the start of treatment that patients (who received prior Ipilimumab/Nivolumab treatment) remained alive, until death from any cause.
Time Frame: Up to 45 months
Population: Treated patients who received prior Ipilimumab/Nivolumab treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 16
months | 7.0 [5.0 to 16.0]

39. Secondary Outcome: 6-month Overall Survival (OS) - Prior Ipilimumab /Nivolumab Treatment
Description: Percentage of patients (previously treated with Ipilimumab/Nivolumab), alive from the start of treatment that patients remain alive, until death from any cause up to 6 months.
Time Frame: Up to 6 months
Population: Treated patients who were previously treated with Ipilimumab/Nivolumab.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 16
percentage of patients | 50 [25 to 71]

40. Secondary Outcome: 12-month Overall Survival (OS) - Prior Ipilimumab / Nivolumab Treatment
Description: Percentage of patients (previously treated with Ipilimumab/Nivolumab), alive from the start of treatment that patients remain alive, until death from any cause up to 12 months.
Time Frame: Up to 12 months
Population: Treated patients who were previously treated with Ipilimumab/Nivolumab.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 16
percentage of patients | 31 [11 to 54]

41. Secondary Outcome: 24-month Overall Survival (OS) - Prior Ipilimumab / Nivolumab Treatment
Description: Percentage of patients (previously treated with Ipilimumab/Nivolumab), alive from the start of treatment that patients remain alive, until death from any cause up to 24 months.
Time Frame: Up to 24 months
Population: Treated patients who were previously treated with Ipilimumab /Nivolumab.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 16
percentage of patients | 19 [5 to 40]

42. Secondary Outcome: Overall Survival (OS) - no Prior Ipilimumab / Nivolumab Treatment
Description: The median number of months from the start of treatment that patients (who did not receive prior Ipilimumab /Nivolumab treatment) remained alive, until death from any cause.
Time Frame: Up to 45 months
Population: Treated patients who do not receive prior Ipilimumab /Nivolumab treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 15
months | 11.0 [7.0 to 23.0]

43. Secondary Outcome: 6-month Overall Survival (OS) - no Prior Ipilimumab /Nivolumab Treatment
Description: Percentage of patients (not previously treated with Ipilimumab /Nivolumab), alive from the start of treatment that patients remain alive, until death from any cause up to 6 months.
Time Frame: Up to 6 months
Population: Treated patients who were not previously treated with Ipilimumab/Nivolumab.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 15
percentage of patients | 93 [61 to 99]

44. Secondary Outcome: 12-month Overall Survival (OS) - no Prior Ipilimumab /Nivolumab Treatment
Description: Percentage of patients (not previously treated with Ipilimumab /Nivolumab), alive from the start of treatment that patients remain alive, until death from any cause up to 12 months.
Time Frame: Up to 12 months
Population: Treated patients who were not previously treated with Ipilimumab/Nivolumab.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 15
percentage of patients | 40 [16 to 63]

45. Secondary Outcome: 24-month Overall Survival (OS) - no Prior Ipilimumab /Nivolumab Treatment
Description: Percentage of patients (not previously treated with Ipilimumab/Nivolumab), alive from the start of treatment that patients remain alive, until death from any cause up to 24 months.
Time Frame: Up to 24 months
Population: Treated patients who were not previously treated with Ipilimumab/Nivolumab.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 15
percentage of patients | 24 [6 to 48]

46. Secondary Outcome: Overall Survival (OS) - Acral Histology
Description: The median number of months from the start of treatment that patients (with acral histology) remain alive, until death from any cause in patients with acral melanoma histology.
Time Frame: Up to 45 months
Population: Treated patients with acral melanoma histology.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 7
months | 8.00 [2.00 to 11.00]

47. Secondary Outcome: 6-month Overall Survival (OS) - Acral Histology
Description: Percentage of patients with acral melanoma histology that remain alive up to 6 months from start of treatment until death from any cause.
Time Frame: Up to 6 months
Population: Treated patients with acral melanoma histology.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 7
percentage of patients | 57 [17 to 84]

48. Secondary Outcome: 12-month Overall Survival (OS) - Acral Histology
Description: Percentage of patients with acral melanoma histology that remain alive up to 12 months from start of treatment until death from any cause.
Time Frame: Up to 12 months
Population: Treated patients with acral melanoma histology.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 7
percentage of patients | 14 [1 to 46]

49. Secondary Outcome: 24-month Overall Survival (OS) - Acral Histology
Description: Percentage of patients with acral melanoma histology that remain alive up to 24 months from start of treatment until death from any cause.
Time Frame: Up to 24 months
Population: Treated patients with acral melanoma histology.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 7
percentage of patients | 14 [1 to 46]

50. Secondary Outcome: Overall Survival (OS) - Mucosal Histology
Description: The median number of months from the start of treatment that patients remain alive, until death from any cause in patients with mucosal histology.
Time Frame: Up to 45 months
Population: Treated patients with mucosal melanoma histology.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 7
months | 11.00 [2.00 to NA] — Upper bound of 95% CI not reached

51. Secondary Outcome: 6-month Overall Survival (OS) - Mucosal Histology
Description: Percentage of patients with mucosal melanoma histology that remain alive up to 6 months from start of treatment until death from any cause.
Time Frame: Up to 6 months
Population: Treated patients with mucosal melanoma histology.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 7
percentage of patients | 71 [26 to 92]

52. Secondary Outcome: 12-month Overall Survival (OS) - Mucosal Histology
Description: Percentage of patients with mucosal melanoma histology that remain alive up to 12 months from start of treatment until death from any cause.
Time Frame: Up to 12 months
Population: Treated patients with mucosal melanoma histology.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 7
percentage of patients | 43 [10 to 73]

53. Secondary Outcome: 24-month Overall Survival (OS) - Mucosal Histology
Description: Percentage of patients with mucosal melanoma histology that remain alive up to 24 months from start of treatment until death from any cause.
Time Frame: Up to 24 months
Population: Treated patients with mucosal melanoma histology.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 7
percentage of patients | 21 [1 to 59]

54. Secondary Outcome: Overall Survival (OS) - Cutaneous Histology
Description: The median number of months from the start of treatment that patients remain alive, until death from any cause in patients with cutaneous melanoma histology.
Time Frame: Up to 45 months
Population: Treated patients with cutaneous melanoma histology
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 17
months | 11.00 [6.00 to 23.00]

55. Secondary Outcome: 6-month Overall Survival (OS) - Cutaneous Histology
Description: Percentage of patients with cutaneous melanoma histology that remain alive up to 6 months from start of treatment until death from any cause.
Time Frame: Up to 6 months
Population: Treated patients with cutaneous melanoma histology.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 17
percentage of patients | 76 [49 to 90]

56. Secondary Outcome: 12-month Overall Survival (OS) - Cutaneous Histology
Description: Percentage of patients with cutaneous melanoma histology that remain alive up to 12 months from start of treatment until death from any cause.
Time Frame: Up to 12 months
Population: Treated patients with cutaneous melanoma histology.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 17
percentage of patients | 41 [19 to 63]

57. Secondary Outcome: 24-month Overall Survival (OS) - Cutaneous Histology
Description: Percentage of patients with cutaneous melanoma histology that remain alive up to 24 months from start of treatment until death from any cause.
Time Frame: Up to 24 months
Population: Treated patients with cutaneous melanoma histology.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 17
percentage of patients | 24 [7 to 45]

58. Secondary Outcome: Overall Survival (OS) - Prior Lines of Therapy >3
Description: The median number of months from the start of treatment that patients with greater than 3 prior lines of treatment remain alive, until death from any cause.
Time Frame: Up to 45 months
Population: Treated patients who received greater than 3 prior lines of treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 11
months | 8.00 [5.00 to 16.00]

59. Secondary Outcome: 6-month Overall Survival (OS) - Prior Lines of Therapy >3
Description: Percentage of patients (who received > 3 prior lines therapy) alive from the start of treatment that patients remain alive, until death from any cause up to 6 months.
Time Frame: Up to 6 months
Population: Treated patients who received >3 prior lines of therapy.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 11
percentage of patients | 73 [37 to 90]

60. Secondary Outcome: 12-month Overall Survival (OS) - Prior Lines of Therapy >3
Description: Percentage of patients (who received > 3 prior lines therapy) alive from the start of treatment that patients remain alive, until death from any cause up to 12 months.
Time Frame: Up to 12 months
Population: Treated patients who received >3 prior lines of therapy.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 11
percentage of patients | 27 [7 to 54]

61. Secondary Outcome: 24-month Overall Survival (OS) - Prior Lines of Therapy >3
Description: Percentage of patients (who received > 3 prior lines therapy) alive from the start of treatment that patients remain alive, until death from any cause up to 24 months.
Time Frame: Up to 24 months
Population: Treated patients who received >3 prior lines of therapy.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 11
percentage of patients | 18 [3 to 44]

62. Secondary Outcome: Overall Survival (OS) - Prior Lines of Therapy <=3
Description: The median number of months from the start of treatment that patients who received 3 or less prior lines of treatment remain alive, until death from any cause.
Time Frame: Up to 45 months
Population: Treated patients who received greater than 3 prior lines of treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 20
months | 11.00 [5.00 to 18.00]

63. Secondary Outcome: 6-month Overall Survival (OS) - Prior Lines of Therapy <=3
Description: Percentage of patients (who received <=3 prior lines therapy) alive from the start of treatment that patients remain alive, until death from any cause up to 6 months.
Time Frame: Up to 6 months
Population: Treated patients who received <=3 prior lines of therapy.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 20
percentage of patients | 70 [45 to 85]

64. Secondary Outcome: 12-month Overall Survival (OS) - Prior Lines of Therapy <=3
Description: Percentage of patients (who received <=3 prior lines therapy) alive from the start of treatment that patients remain alive, until death from any cause up to 12 months.
Time Frame: Up to 12 months
Population: Treated patients who received <=3 prior lines of therapy.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 20
percentage of patients | 40 [19 to 60]

65. Secondary Outcome: 24-month Overall Survival (OS) - Prior Lines of Therapy <=3
Description: Percentage of patients (who received <=3 prior lines therapy) alive from the start of treatment that patients remain alive, until death from any cause up to 24 months.
Time Frame: Up to 24 months
Population: Treated patients who received <=3 prior lines of therapy.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 20
percentage of patients | 23 [7 to 43]

66. Secondary Outcome: Overall Survival (OS) - Overall Cohort - Primary IO Resistance
Description: The median number of months from the start of treatment that patients with Primary IO resistance remain alive, until death from any cause.
Time Frame: Up to 45 months
Population: Treated patients with Primary IO resistance.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 15
months | 7.00 [3.00 to 16.00]

67. Secondary Outcome: 6-month Overall Survival (OS) - Primary IO Resistance
Description: Percentage of patients (Primary IO resistance) alive from the start of treatment that patients remain alive, until death from any cause up to 6 months.
Time Frame: Up to 6 months
Population: Treated patients with Primary IO resistance.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 15
percentage of patients | 53 [26 to 74]

68. Secondary Outcome: 12-month Overall Survival (OS) - Primary IO Resistance
Description: Percentage of patients (Primary IO resistance) alive from the start of treatment that patients remain alive, until death from any cause up to 12 months.
Time Frame: Up to 12 months
Population: Treated patients with Primary IO resistance.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 15
percentage of patients | 40 [16 to 63]

69. Secondary Outcome: 24-month Overall Survival (OS) - Primary IO Resistance
Description: Percentage of patients (Primary IO resistance) alive from the start of treatment that patients remain alive, until death from any cause up to 24 months.
Time Frame: Up to 24 months
Population: Treated patients with Primary IO resistance.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 14
percentage of patients | 24 [6 to 48]

70. Secondary Outcome: Overall Survival (OS) - Overall Cohort - Secondary IO Resistance
Description: The median number of months from the start of treatment that patients with Secondary IO resistance remain alive, until death from any cause.
Time Frame: Up to 45 months
Population: Treated patients with Primary IO resistance.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 16
months | 11.00 [8.00 to 18.00]

71. Secondary Outcome: 6-month Overall Survival (OS) - Secondary IO Resistance
Description: Percentage of patients with Secondary IO resistance alive from the start of treatment that patients remain alive, until death from any cause up to 6 months.
Time Frame: Up to 6 months
Population: Treated patients with Secondary IO resistance.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 16
percentage of patients | 88 [59 to 97]

72. Secondary Outcome: 12-month Overall Survival (OS) - Secondary IO Resistance
Description: Percentage of patients with Secondary IO resistance alive from the start of treatment that patients remain alive, until death from any cause up to 12 months.
Time Frame: Up to 12 months
Population: Treated patients with Secondary IO resistance.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 16
percentage of patients | 31 [11 to 54]

73. Secondary Outcome: 24-month Overall Survival (OS) - Secondary IO Resistance
Description: Percentage of patients with Secondary IO resistance alive from the start of treatment that patients remain alive, until death from any cause up to 24 months.
Time Frame: Up to 24 months
Population: Treated patients with Secondary IO resistance.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 16
percentage of patients | 19 [5 to 40]

74. Secondary Outcome: Progression-free Survival (PFS) - Overall Cohort
Description: The median time measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression), whichever occurs first, with progression defined by RECIST v 1.1. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Time Frame: Up to 4 years and 3 months
Population: Treated patients who were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 30
months | 3.00 [3.00 to 5.00]

75. Secondary Outcome: 6-month Progression-free Survival (PFS)
Description: The percentage of patients who do not experience documented progression, or death (in the absence of progression), whichever occurs first, within 6 months start of treatment. Per RECIST v 1.1. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Time Frame: Up to 6 months
Population: Treated patients who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 30
percentage of patients | 21 [9 to 37]

76. Secondary Outcome: 12-month Progression-free Survival (PFS)
Description: The percentage of patients who do not experience documented progression, or death (in the absence of progression), whichever occurs first, within 12 months start of treatment. Per RECIST v 1.1. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Time Frame: Up to 12 months
Population: Treated patients who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 30
percentage of patients | 11 [3 to 25]

77. Secondary Outcome: 24-month Progression-free Survival (PFS)
Description: The percentage of patients who do not experience documented progression, or death (in the absence of progression), whichever occurs first, within 24 months start of treatment. Per RECIST v 1.1. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Time Frame: Up to 24 months
Population: Treated patients who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 29
percentage of patients | 0 [0 to 0]

78. Secondary Outcome: Progression-free Survival (PFS) - Prior Ipilimumab / Nivolumab Treatment
Description: as for outcome 74
Time Frame: Up to 4 years and 3 months
Population: Treated patients who were previously treated with Ipilimumab/Nivolumab and were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 16
months | 4.00 [3.00 to 6.00]

79. Secondary Outcome: 6-month Progression-free Survival (PFS) - Prior Ipilimumab / Nivolumab Treatment
Description: The percentage of patients (previously treated with Ipilimumab/Nivolumab) who do not experience documented progression, or death (in the absence of progression), whichever occurs first, within 6 months start of treatment. Per RECIST v 1.1. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Time Frame: Up to 6 months
Population: Treated patients who were previously treated with Ipilimumab /Nivolumab and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 16
percentage of patients | 19 [5 to 40]

80. Secondary Outcome: 12-month Progression-free Survival (PFS) - Prior Ipilimumab / Nivolumab Treatment
Description: The percentage of patients (previously treated with Ipilimumab / Nivolumab) who do not experience documented progression, or death (in the absence of progression), whichever occurs first, within 12 months start of treatment. Per RECIST v 1.1. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Time Frame: Up to 12 months
Population: Treated patients who were previously treated with Ipilimumab /Nivolumab and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 16
percentage of patients | 13 [2 to 33]

81. Secondary Outcome: 24-month Progression-free Survival (PFS) - Prior Ipilimumab / Nivolumab Treatment
Description: The percentage of patients (previously treated with Ipilimumab/Nivolumab) who do not experience documented progression, or death (in the absence of progression), whichever occurs first, within 24 months start of treatment. Per RECIST v 1.1. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Time Frame: Up to 24 months
Population: Treated patients who were previously treated with Ipilimumab /Nivolumab and were evaluable for radiologic response.
Measure: Number; unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 15
percentage of patients | 0

82. Secondary Outcome: Progression-free Survival (PFS) - no Prior Ipilimumab /Nivolumab Treatment
Description: as for outcome 74
Time Frame: Up to 4 years and 3 months
Population: Treated patients who were not previously treated with Ipilimumab /Nivolumab and were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 14
months | 3.00 [2.00 to 4.00]

83. Secondary Outcome: 6-month Progression-free Survival (PFS) - no Prior Ipilimumab/Nivolumab Treatment
Description: The percentage of patients (not previously treated with Ipilimumab /Nivolumab) who do not experience documented progression, or death (in the absence of progression), whichever occurs first, within 6 months start of treatment. Per RECIST v 1.1. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Time Frame: Up to 6 months
Population: Treated patients who were not previously treated with Ipilimumab /Nivolumab and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 14
percentage of patients | 27 [8 to 50]

84. Secondary Outcome: 12-month Progression-free Survival (PFS) - no Prior Ipilimumab / Nivolumab Treatment
Description: The percentage of patients (not previously treated with Ipilimumab /Nivolumab) who do not experience documented progression, or death (in the absence of progression), whichever occurs first, within 12 months start of treatment. Per RECIST v 1.1. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Time Frame: Up to 12 months
Population: Treated patients who were not previously treated with Ipilimumab /Nivolumab and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 14
percentage of patients | 9 [1 to 32]

85. Secondary Outcome: 24-month Progression-free Survival (PFS) - no Prior Ipilimumab /Nivolumab Treatment
Description: The percentage of patients (not previously treated with Ipilimumab /Nivolumab) who do not experience documented progression, or death (in the absence of progression), whichever occurs first, within 24 months start of treatment. Per RECIST v 1.1. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Time Frame: Up to 24 months
Population: Treated patients who were not previously treated with Ipilimumab /Nivolumab and were evaluable for radiologic response.
Measure: Number; unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 14
percentage of patients | 0

86. Secondary Outcome: Progression-free Survival (PFS) - Overall Cohort - Mucosal Histology
Description: The median time measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression), whichever occurs first, with progression defined by RECIST v 1.1. in patients with mucosal histology. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Time Frame: Up to 4 years and 3 months
Population: Treated patients with mucosal histology who were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 6
months | 3.00 [1.00 to NA] — Upper bound of 95% CI not reached

87. Secondary Outcome: 6-month Progression-free Survival (PFS) - Mucosal Histology
Description: The percentage of patients (with mucosal histology) who do not experience documented progression, or death (in the absence of progression), whichever occurs first, within 6 months start of treatment. Per RECIST v 1.1. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Time Frame: Up to 6 months
Population: Treated patients with mucosal histology and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 6
percentage of patients | 29 [4 to 61]

88. Secondary Outcome: 12-month Progression-free Survival (PFS) - Mucosal Histology
Description: The percentage of patients (with mucosal histology) who do not experience documented progression, or death (in the absence of progression), whichever occurs first, within 12 months start of treatment. Per RECIST v 1.1. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Time Frame: Up to 12 months
Population: Treated patients with mucosal histology and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 6
percentage of patients | 0 [NA to NA] — 95% CI not reached

89. Secondary Outcome: 24-month Progression-free Survival (PFS) - Mucosal Histology
Description: The percentage of patients (with mucosal histology) who do not experience documented progression, or death (in the absence of progression), whichever occurs first, within 24 months start of treatment. Per RECIST v 1.1. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Time Frame: Up to 24 months
Population: Treated patients with mucosal histology and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 6
percentage of patients | 0 [NA to NA] — 95% CI not reached

90. Secondary Outcome: Progression-free Survival (PFS) - Overall Cohort - Cutaneous Histology
Description: as for outcome 86
Time Frame: Up to 4 years and 3 months
Population: Treated patients with cutaneous histology who were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 17
months | 3.00 [2.00 to 6.00]

91. Secondary Outcome: 6-month Progression-free Survival (PFS) - Cutaneous Histology
Description: The percentage of patients (with cutaneous histology) who do not experience documented progression, or death (in the absence of progression), whichever occurs first, within 6 months start of treatment. Per RECIST v 1.1. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Time Frame: Up to 6 months
Population: Treated patients with cutaneous histology and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 17
percentage of patients | 18 [4 to 38]

92. Secondary Outcome: 12-month Progression-free Survival (PFS) - Cutaneous Histology
Description: as for outcome 91
Time Frame: Up to 12 months
Population: Treated patients with cutaneous histology and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 17
percentage of patients | 18 [4 to 38]

93. Secondary Outcome: 24-month Progression-free Survival (PFS) - Cutaneous Histology
Description: as for outcome 91
Time Frame: Up to 24 months
Population: Treated patients with cutaneous histology and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 16
percentage of patients | 0 [NA to NA] — 95% CI not reached

94. Secondary Outcome: Progression-free Survival (PFS) - Overall Cohort - Acral Histology
Description: as for outcome 86
Time Frame: Up to 4 years and 3 months
Population: Treated patients with acral histology who were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 7
months | 4.00 [0.00 to 8.00]

95. Secondary Outcome: 6-month Progression-free Survival (PFS) - Acral Histology
Description: The percentage of patients (with acral histology) who do not experience documented progression, or death (in the absence of progression), whichever occurs first, within 6 months start of treatment. Per RECIST v 1.1. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Time Frame: Up to 6 months
Population: Treated patients with acral histology and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 7
percentage of patients | 29 [4 to 61]

96. Secondary Outcome: 12-month Progression-free Survival (PFS) - Acral Histology
Description: as for outcome 95
Time Frame: Up to 12 months
Population: Treated patients with acral histology and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 7
percentage of patients | 0 [NA to NA] — 95% CI not reached

97. Secondary Outcome: 24-month Progression-free Survival (PFS) - Acral Histology
Description: as for outcome 95
Time Frame: Up to 24 months
Population: Treated patients with acral histology and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 7
percentage of patients | 0 [NA to NA] — 95% CI not reached

98. Secondary Outcome: Progression-free Survival (PFS) - Overall Cohort - Prior Lines <= 3
Description: as for outcome 86
Time Frame: Up to 4 years and 3 months
Population: Treated patients who received prior lines <= 3 and who were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 19
months | 3.50 [2.00 to 6.00]

99. Secondary Outcome: 6-month Progression-free Survival (PFS) - Prior Lines <= 3
Description: as for outcome 75
Time Frame: Up to 6 months
Population: Treated patients who received <=3 prior lines of therapy and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 19
percentage of patients | 28 [11 to 49]

100. Secondary Outcome: 12-month Progression-free Survival (PFS) - Prior Lines <= 3
Description: as for outcome 76
Time Frame: Up to 12 months
Population: Treated patients who received <=3 prior lines of therapy and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 19
percentage of patients | 11 [2 to 30]

101. Secondary Outcome: 24-month Progression-free Survival (PFS) - Prior Lines <= 3
Description: as for outcome 77
Time Frame: Up to 24 months
Population: Treated patients who received <=3 prior lines of therapy and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 19
percentage of patients | 0 [NA to NA] — 95% CI not reached

102. Secondary Outcome: Progression-free Survival (PFS) - Overall Cohort - Prior Lines >3
Description: as for outcome 86
Time Frame: Up to 4 years and 3 months
Population: Treated patients who received >3 prior lines and who were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 11
months | 3.00 [2.00 to 4.00]

103. Secondary Outcome: 6-month Progression-free Survival (PFS) - Prior Lines > 3
Description: as for outcome 75
Time Frame: Up to 6 months
Population: Treated patients who received >3 prior lines of therapy and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 11
percentage of patients | 9 [1 to 33]

104. Secondary Outcome: 12-month Progression-free Survival (PFS) - Prior Lines > 3
Description: as for outcome 76
Time Frame: Up to 12 months
Population: Treated patients who received >3 prior lines of therapy and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 11
percentage of patients | 9 [1 to 33]

105. Secondary Outcome: 24-month Progression-free Survival (PFS) - Prior Lines > 3
Description: as for outcome 77
Time Frame: Up to 24 months
Population: Treated patients who received >3 prior lines of therapy and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 11
percentage of patients | 0 [NA to NA] — 95% CI not reached

106. Secondary Outcome: Duration of Response (DoR) - Overall Cohort
Description: Median number of months from the first confirmed response (CR/PR) to date of the first progression or death from any cause. Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR) is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 4 years and 3 months
Population: Treated patients who were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 31
months | 8.00 [4.00 to NA] — Upper bound of 95% CI not reached

107. Secondary Outcome: 6-month Duration of Response (DoR) - Overall Cohort
Description: Percentage of patients whose Complete Response (CR) or Partial Response (PR) remains as such at 6 months from date of first confirmed response. Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR) is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 6 months
Population: Treated patients who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 3
percentage of patients | 67 [5 to 95]

108. Secondary Outcome: 12-month Duration of Response (DoR) - Overall Cohort
Description: Percentage of patients whose Complete Response (CR) or Partial Response (PR) remains as such at 12 months from date of first confirmed response. Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR) is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 12 months
Population: Treated patients who were evaluable for radiologic response.
Measure: Number; unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 3
percentage of patients | 0

109. Secondary Outcome: 24-month Duration of Response (DoR) - Overall Cohort
Description: Percentage of patients whose Complete Response (CR) or Partial Response (PR) remains as such at 24 months from date of first confirmed response. Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR) is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 24 months
Population: Treated patients who were evaluable for radiologic response.
Measure: Number; unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 3
percentage of patients | 0

110. Secondary Outcome: Duration of Response (DoR) - Prior Ipilimumab / Nivolumab Treatment
Description: as for outcome 106
Time Frame: Up to 4 years and 3 months
Population: Treated patients who received prior Ipilimumab/Nivolumab treatment were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 1
months | 0 [NA to NA] — 95% CI not reached

111. Secondary Outcome: 6-month Duration of Response (DoR) - Prior Ipilimumab / Nivolumab Treatment
Description: as for outcome 107
Time Frame: Up to 6 months
Population: Treated patients who received prior Ipilimumab/Nivolumab treatment were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 1
percentage of patients | 0 [NA to NA] — 95% CI not reached

112. Secondary Outcome: 12-month Duration of Response (DoR) - Prior Ipilimumab / Nivolumab Treatment
Description: as for outcome 108
Time Frame: Up to 12 months
Population: Treated patients who received prior Ipilimumab/Nivolumab treatment were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 1
percentage of patients | 0 [NA to NA] — 95% CI not reached

113. Secondary Outcome: 24-month Duration of Response (DoR) - Prior Ipilimumab / Nivolumab Treatment
Description: as for outcome 109
Time Frame: Up to 24 months
Population: Treated patients who received prior Ipilimumab/Nivolumab treatment were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 1
percentage of patients | 0 [NA to NA] — 95% CI not reached

114. Secondary Outcome: Duration of Response (DoR) - no Prior Ipilimumab / Nivolumab Treatment
Description: as for outcome 106
Time Frame: Up to 4 years and 3 months
Population: Treated patients who did not receive prior Ipilimumab / Nivolumab treatment and were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 2
months | 8.50 [8.00 to NA] — Upper bound of 95% CI not reached

115. Secondary Outcome: 6-month Duration of Response (DoR) - no Prior Ipilimumab / Nivolumab Treatment
Description: as for outcome 107
Time Frame: Up to 6 months
Population: Treated patients who did not received prior Ipilimumab/Nivolumab treatment were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 2
percentage of patients | 100.00 [100 to 100]

116. Secondary Outcome: 12-month Duration of Response (DoR) - no Prior Ipilimumab / Nivolumab Treatment
Description: as for outcome 108
Time Frame: Up to 12 months
Population: Treated patients who did not received prior Ipilimumab/Nivolumab treatment were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 2
percentage of patients | 0 [NA to NA] — 95% CI not reached

117. Secondary Outcome: 24-month Duration of Response (DoR) - no Prior Ipilimumab / Nivolumab Treatment
Description: as for outcome 109
Time Frame: Up to 24 months
Population: Treated patients who did not received prior Ipilimumab/Nivolumab treatment were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 2
percentage of patients | 0 [NA to NA] — 95% CI not reached

118. Secondary Outcome: Duration of Response (DoR) - Acral Histology
Description: as for outcome 106
Time Frame: Up to 4 years and 3 months
Population: Treated patients with acral histology who were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 1
months | 9.0 [NA to NA] — 95% CI not reached

119. Secondary Outcome: 6-month Duration of Response (DoR) - Acral Histology
Description: as for outcome 107
Time Frame: Up to 6 months
Population: Treated patients with acral histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 1
percentage of patients | 100 [NA to NA] — 95% CI Not Available

120. Secondary Outcome: 12-month Duration of Response (DoR) - Acral Histology
Description: as for outcome 108
Time Frame: Up to 12 months
Population: Treated patients with acral histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 1
percentage of patients | 0 [NA to NA] — 95% CI not reached

121. Secondary Outcome: 24-month Duration of Response (DoR) - Acral Histology
Description: as for outcome 109
Time Frame: Up to 24 months
Population: Treated patients with acral histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 1
percentage of patients | 0 [NA to NA] — 95% CI not reached

122. Secondary Outcome: Duration of Response (DoR) - Mucosal Histology
Description: as for outcome 106
Time Frame: Up to 4 years and 3 months
Population: Treated patients with mucosal histology who were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 1
months | 8.00 [NA to NA] — 95% CI not reached

123. Secondary Outcome: 6-month Duration of Response (DoR) - Mucosal Histology
Description: as for outcome 107
Time Frame: Up to 6 months
Population: Treated patients with mucosal histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 1
percentage of patients | 100 [NA to NA] — 95% CI Not Available

124. Secondary Outcome: 12-month Duration of Response (DoR) - Mucosal Histology
Description: as for outcome 108
Time Frame: Up to 12 months
Population: Treated patients with mucosal histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 1
percentage of patients | 0 [NA to NA] — 95% CI not reached

125. Secondary Outcome: 24-month Duration of Response (DoR) - Mucosal Histology
Description: as for outcome 109
Time Frame: Up to 24 months
Population: Treated patients with mucosal histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 1
percentage of patients | 0 [NA to NA] — 95% CI not reached

126. Secondary Outcome: Duration of Response (DoR) - Cutaneous Histology
Description: as for outcome 106
Time Frame: Up to 4 years and 3 months
Population: Treated patients with cutaneous histology who were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 1
months | 4.00 [NA to NA] — 95% CI not reached

127. Secondary Outcome: 6-month Duration of Response (DoR) - Cutaneous Histology
Description: as for outcome 107
Time Frame: Up to 6 months
Population: Treated patients with cutaneous histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 1
percentage of patients | 0 [NA to NA] — 95% CI not reached

128. Secondary Outcome: 12-month Duration of Response (DoR) - Cutaneous Histology
Description: as for outcome 108
Time Frame: Up to 12 months
Population: Treated patients with cutaneous histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 1
percentage of patients | 0 [NA to NA] — 95% CI not reached

129. Secondary Outcome: 24-month Duration of Response (DoR) - Cutaneous Histology
Description: as for outcome 109
Time Frame: Up to 24 months
Population: Treated patients with cutaneous histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 1
percentage of patients | 0 [NA to NA] — 95% CI not reached

130. Secondary Outcome: Duration of Disease Control (DoDC) - Overall Cohort
Description: Median number of months from the date of first disease control (i.e. complete response [CR], partial response [PR], and stable disease [SD]) to progression [PD]. Per RECIST v1.1, (CR) = disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. (PR) = at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. (SD) = neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study. PD = at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Time Frame: Up to 4 years and 3 months
Population: Treated patients who were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 13
months | 4.00 [2.00 to 8.00]

131. Secondary Outcome: 6-month Duration of Disease Control (DoDC) - Overall Cohort
Description: Percentage of patients with first disease control (i.e. complete response [CR], partial response [PR], and stable disease [SD]) to progression [PD]. Per RECIST v1.1, (CR) = disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. (PR) = at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. (SD) = neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study. PD = at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Time Frame: Up to 6 months
Population: Treated patients who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 13
percentage of patients | 39 [14 to 63]

132. Secondary Outcome: 12-month Duration of Disease Control (DoDC) - Overall Cohort
Description: as for outcome 131
Time Frame: Up to 12 months
Population: Treated patients who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 13
percentage of patients | 15 [2 to 39]

133. Secondary Outcome: 24-month Duration of Disease Control (DoDC) - Overall Cohort
Description: as for outcome 131
Time Frame: Up to 24 months
Population: Treated patients who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 12
percentage of patients | 0 [NA to NA] — 95% CI not reached

134. Secondary Outcome: Duration of Disease Control (DoDC) - Prior Ipilimumab / Nivolumab Treatment
Description: as for outcome 130
Time Frame: Up to 4 years and 3 months
Population: Treated patients who received prior Ipilimumab / Nivolumab treatment and were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 9
months | 3.00 [2.00 to 15.00]

135. Secondary Outcome: 6-month Duration of Disease Control (DoDC) - Prior Ipilimumab / Nivolumab Treatment
Description: as for outcome 131
Time Frame: Up to 6 months
Population: Treated patients who received Prior Ipilimumab / Nivolumab Treatment and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 9
percentage of patients | 22 [3 to 51]

136. Secondary Outcome: 12-month Duration of Disease Control (DoDC) - Prior Ipilimumab / Nivolumab Treatment
Description: as for outcome 131
Time Frame: Up to 12 months
Population: Treated patients who received Prior Ipilimumab / Nivolumab Treatment and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 9
percentage of patients | 22 [3 to 51]

137. Secondary Outcome: 24-month Duration of Disease Control (DoDC) - Prior Ipilimumab / Nivolumab Treatment
Description: as for outcome 131
Time Frame: Up to 24 months
Population: Treated patients who received Prior Ipilimumab / Nivolumab Treatment and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 9
percentage of patients | 0 [NA to NA] — 95% CI not reached

138. Secondary Outcome: Duration of Disease Control (DoDC) - no Prior Ipilimumab / Nivolumab Treatment
Description: as for outcome 130
Time Frame: Up to 4 years and 3 months
Population: Treated patients who did not received prior Ipilimumab / Nivolumab treatment and were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 4
months | 8.00 [1.00 to NA] — Upper bound of 95% CI not reached

139. Secondary Outcome: 6-month Duration of Disease Control (DoDC) - no Prior Ipilimumab / Nivolumab Treatment
Description: as for outcome 131
Time Frame: Up to 6 months
Population: Treated patients who did not received Prior Ipilimumab / Nivolumab Treatment and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 4
percentage of patients | 80 [20 to 97]

140. Secondary Outcome: 12-month Duration of Disease Control (DoDC) - no Prior Ipilimumab / Nivolumab Treatment
Description: as for outcome 131
Time Frame: Up to 12 months
Population: Treated patients who did not received Prior Ipilimumab / Nivolumab Treatment and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 4
percentage of patients | 0 [NA to NA] — 95% CI not reached

141. Secondary Outcome: 24-month Duration of Disease Control (DoDC) - no Prior Ipilimumab / Nivolumab Treatment
Description: as for outcome 131
Time Frame: Up to 24 months
Population: Treated patients who did not received Prior Ipilimumab / Nivolumab Treatment and were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 4
percentage of patients | 0 [NA to NA] — Upper bound of 95% CI not reached

142. Secondary Outcome: Duration of Disease Control (DoDC) - Acral Histology
Description: as for outcome 130
Time Frame: Up to 4 years and 3 months
Population: Treated patients with acral histology who were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 5
months | 3.00 [2.00 to NA] — Upper bound of 95% CI not reached

143. Secondary Outcome: 6-month Duration of Disease Control (DoDC) - Acral Histology
Description: as for outcome 131
Time Frame: Up to 6 months
Population: Treated patients with acral histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 5
percentage of patients | 20 [1 to 58]

144. Secondary Outcome: 12-month Duration of Disease Control (DoDC) - Acral Histology
Description: as for outcome 131
Time Frame: Up to 12 months
Population: Treated patients with acral histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 5
percentage of patients | 0 [NA to NA] — 95% CI not reached

145. Secondary Outcome: 24-month Duration of Disease Control (DoDC) - Acral Histology
Description: as for outcome 131
Time Frame: Up to 24 months
Population: Treated patients with acral histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 5
percentage of patients | 0 [NA to NA] — 95% CI not reached

146. Secondary Outcome: Duration of Disease Control (DoDC) - Mucosal Histology
Description: as for outcome 130
Time Frame: Up to 4 years and 3 months
Population: Treated patients with mucosal histology who were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 2
months | 8.00 [1.00 to NA] — Upper bound of 95% CI not reached

147. Secondary Outcome: 6-month Duration of Disease Control (DoDC) - Mucosal Histology
Description: as for outcome 131
Time Frame: Up to 6 months
Population: Treated patients with mucosal histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 2
percentage of patients | 67 [5 to 95]

148. Secondary Outcome: 12-month Duration of Disease Control (DoDC) - Mucosal Histology
Description: as for outcome 131
Time Frame: Up to 12 months
Population: Treated patients with mucosal histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 2
percentage of patients | 0 [NA to NA] — 95% CI not reached

149. Secondary Outcome: 24-month Duration of Disease Control (DoDC) - Mucosal Histology
Description: as for outcome 131
Time Frame: Up to 24 months
Population: Treated patients with mucosal histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 2
percentage of patients | 0 [NA to NA] — 95% CI not reached

150. Secondary Outcome: Duration of Disease Control (DoDC) - Cutaneous Histology
Description: as for outcome 130
Time Frame: Up to 4 years and 3 months
Population: Treated patients with cutaneous histology who were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 6
months | 6.00 [2.00 to NA] — Upper bound of 95% CI nor reached

151. Secondary Outcome: 6-month Duration of Disease Control (DoDC) - Cutaneous Histology
Description: as for outcome 131
Time Frame: Up to 6 months
Population: Treated patients with cutaneous histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 6
percentage of patients | 50 [11 to 80]

152. Secondary Outcome: 12-month Duration of Disease Control (DoDC) - Cutaneous Histology
Description: as for outcome 131
Time Frame: Up to 12 months
Population: Treated patients with cutaneous histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 6
percentage of patients | 33 [5 to 68]

153. Secondary Outcome: 24-month Duration of Disease Control (DoDC) - Cutaneous Histology
Description: as for outcome 131
Time Frame: Up to 24 months
Population: Treated patients with cutaneous histology who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 5
percentage of patients | 0 [NA to NA] — 95% CI not reached

154. Secondary Outcome: Duration of Disease Control (DoDC) - Prior Lines > 3
Description: as for outcome 130
Time Frame: Up to 4 years and 3 months
Population: Treated patients who received >3 prior lines of therapy and were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 4
months | 2.00 [2.00 to NA] — Upper bound of 95% CI not reached

155. Secondary Outcome: 6-month Duration of Disease Control (DoDC) - Prior Lines > 3
Description: as for outcome 131
Time Frame: Up to 6 months
Population: Treated patients who received > 3 prior lines of therapy and who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 4
percentage of patients | 25 [1 to 67]

156. Secondary Outcome: 12-month Duration of Disease Control (DoDC) - Prior Lines > 3
Description: as for outcome 131
Time Frame: Up to 12 months
Population: Treated patients who received > 3 prior lines of therapy and who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 4
percentage of patients | 25 [1 to 67]

157. Secondary Outcome: 24-month Duration of Disease Control (DoDC) - Prior Lines > 3
Description: as for outcome 131
Time Frame: Up to 24 months
Population: Treated patients who received > 3 prior lines of therapy and who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 3
percentage of patients | 0 [NA to NA] — 95% CI not reached

158. Secondary Outcome: Duration of Disease Control (DoDC) - Prior Lines <= 3
Description: as for outcome 130
Time Frame: Up to 4 years and 3 months
Population: Treated patients who received <= 3 prior lines of therapy and were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 9
months | 5.00 [1.00 to 9.00]

159. Secondary Outcome: 6-month Duration of Disease Control (DoDC) - Prior Lines <= 3
Description: as for outcome 131
Time Frame: Up to 6 months
Population: Treated patients who received <= 3 prior lines of therapy and who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 9
percentage of patients | 45 [14 to 72]

160. Secondary Outcome: 12-month Duration of Disease Control (DoDC) - Prior Lines <= 3
Description: as for outcome 131
Time Frame: Up to 12 months
Population: Treated patients who received <= 3 prior lines of therapy and who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 9
percentage of patients | 11 [1 to 39]

161. Secondary Outcome: 24-month Duration of Disease Control (DoDC) - Prior Lines <= 3
Description: as for outcome 131
Time Frame: Up to 24 months
Population: Treated patients who received <= 3 prior lines of therapy and who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 9
percentage of patients | 0 [NA to NA] — 95% CI not reached

162. Secondary Outcome: Duration of Disease Control (DoDC) - Overall Cohort - Primary IO Resistance
Description: as for outcome 130
Time Frame: Up to 4 years and 3 months
Population: Treated patients with primary IO resistance who were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 7
months | 3.00 [2.00 to 8.00]

163. Secondary Outcome: 6-month Duration of Disease Control (DoDC) - Primary IO Resistance
Description: as for outcome 131
Time Frame: Up to 6 months
Population: Treated patients with primary IO resistance who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 7
percentage of patients | 29 [4 to 61]

164. Secondary Outcome: 12-month Duration of Disease Control (DoDC) - Primary IO Resistance
Description: as for outcome 131
Time Frame: Up to 12 months
Population: Treated patients with primary IO resistance who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 7
percentage of patients | 14 [1 to 46]

165. Secondary Outcome: 24-month Duration of Disease Control (DoDC) - Primary IO Resistance
Description: as for outcome 131
Time Frame: Up to 24 months
Population: Treated patients with primary IO resistance who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 6
percentage of patients | 0 [NA to NA] — 95% CI not reached

166. Secondary Outcome: Duration of Disease Control (DoDC) - Overall Cohort - Secondary IO Resistance
Description: as for outcome 130
Time Frame: Up to 4 years and 3 months
Population: Treated patients with Secondary IO resistance who were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 6
months | 6.00 [1.00 to NA] — Upper bound of 95% CI not reached

167. Secondary Outcome: 6-month Duration of Disease Control (DoDC) - Secondary IO Resistance
Description: as for outcome 131
Time Frame: Up to 6 months
Population: Treated patients with Secondary IO resistance who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 6
percentage of patients | 50 [11 to 80]

168. Secondary Outcome: 12-month Duration of Disease Control (DoDC) - Secondary IO Resistance
Description: as for outcome 131
Time Frame: Up to 12 months
Population: Treated patients with Secondary IO resistance who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 6
percentage of patients | 17 [1 to 52]

169. Secondary Outcome: 24-month Duration of Disease Control (DoDC) - Secondary IO Resistance
Description: as for outcome 131
Time Frame: Up to 24 months
Population: Treated patients with Secondary IO resistance who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 6
percentage of patients | 0 [NA to NA] — 95% CI not reached

170. Secondary Outcome: Grade 3 or Greater Adverse Events Possibly, Probably or Definitely Related to Study Treatment
Description: Adverse Events determined to be possibly, probably or definitely related to study treatment SAEs are defined as grade 3 and higher toxicity events that are attributable to the study combination therapy. Evaluated by NCI Common Terminology for Adverse Events (CTCAE v5.0).
Time Frame: Up to 28 days after discontinuation of study treatment (up to 24 months)
Population: Treated patients who experienced an SAE >= grade 3
Measure: Number; unit: participants
Arm/Group | Nivolumab Plus Axitinib
Number analyzed (Participants) | 10
participants
  Diarrhea | 1
  Lower gastrointestinal hemorrhage | 1
  Chills | 1
  Fatigue | 1
  dacryocystitis | 1
  Wound complication | 1
  Alkaline phosphatase increased | 1
  Hematuria | 1
  Pneumonitis | 1
  Rash maculo-papular | 1

ADVERSE EVENTS:
Time Frame: Adverse events data collected for to up to 28 days after discontinuation of study treatment (up to 24 months) for individual patients. All-Cause Mortality data were collected for up to up to 4 years and 3 months
Arm/Group | Nivolumab Plus Axitinib
All-Cause Mortality (participants affected / at risk) | 26/31
Serious Adverse Events (participants affected / at risk) | 15/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab Plus Axitinib (N=31)
Heart failure (Cardiac disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 1
Flu like symptoms (General disorders) | 1
Infections and infestations - Other, specify: dacryocystitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Wound complication (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify: Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Paresthesia (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
left brachial and axillary ulnar and radial thrombectomies (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab Plus Axitinib (N=31)
Anemia (Blood and lymphatic system disorders) | 16
Blood and lymphatic system disorders - Other, specify: Eosinophilia (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, specify: eosinophilia (Blood and lymphatic system disorders) | 3
Blood and lymphatic system disorders - Other, specify: splenic infarct (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 2
Heart failure (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 4
Sinus tachycardia (Cardiac disorders) | 1
Middle ear inflammation (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Blurred vision (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 4
Anal fistula (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 9
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: constipation (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: diarrhea (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify: dry heaving (int) (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 8
Oral pain (Gastrointestinal disorders) | 5
Rectal mucositis (Gastrointestinal disorders) | 1
Rectal pain (Gastrointestinal disorders) | 2
Stomach pain (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Chills (General disorders) | 1
Edema limbs (General disorders) | 3
Facial pain (General disorders) | 1
Fatigue (General disorders) | 17
Fever (General disorders) | 1
Flu like symptoms (General disorders) | 2
Gait disturbance (General disorders) | 2
General disorders and administration site conditions - Other, specify: Edema (General disorders) | 1
General disorders and administration site conditions - Other, specify: Fever (General disorders) | 1
General disorders and administration site conditions - Other, specify: Pain (General disorders) | 2
Infusion related reaction (General disorders) | 1
Injection site reaction (General disorders) | 1
Pain (General disorders) | 6
Infections and infestations - Other, specify: Chest Wall Infection (Infections and infestations) | 1
Infections and infestations - Other, specify: Covid-19 (Infections and infestations) | 1
Infections and infestations - Other, specify: Lyme's disease (Infections and infestations) | 1
Infections and infestations - Other, specify: dacryocystitis (Infections and infestations) | 1
Infections and infestations - Other, specify: skin infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Bruising (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Wound complication (Injury, poisoning and procedural complications) | 2
Activated partial thromboplastin time prolonged (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 7
Alkaline phosphatase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 8
Blood bicarbonate decreased (Investigations) | 1
Blood bilirubin increased (Investigations) | 4
Blood lactate dehydrogenase increased (Investigations) | 14
CPK increased (Investigations) | 1
Creatinine increased (Investigations) | 7
Hemoglobin increased (Investigations) | 3
INR increased (Investigations) | 3
Investigations - Other, specify: Blood Urea Nitrogen Increased (Investigations) | 1
Investigations - Other, specify: Free T4 decreased (Investigations) | 1
Investigations - Other, specify: Increased CRP (Investigations) | 1
Investigations - Other, specify: Increased D Dimer (Investigations) | 1
Investigations - Other, specify: T3 Decreased (Investigations) | 1
Investigations - Other, specify: TSH increased (Investigations) | 1
Investigations - Other, specify: blood CO2 increased (Investigations) | 1
Investigations - Other, specify: increased urine ketones (Investigations) | 1
Investigations - Other, specify: urine microalbumin increased (Investigations) | 1
Investigations - Other, specify: urine specific gravity increased (Investigations) | 1
Lipase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 10
Lymphocyte count increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 6
Thyroid stimulating hormone increased (Investigations) | 11
Weight loss (Investigations) | 6
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 11
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 9
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 11
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 22
Hypophosphatemia (Metabolism and nutrition disorders) | 6
Obesity (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify: Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Paresthesia (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Confusion (Psychiatric disorders) | 4
Delirium (Psychiatric disorders) | 1
Hallucinations (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 6
Proteinuria (Renal and urinary disorders) | 7
Urinary frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Prostatic obstruction (Reproductive system and breast disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify: Septal Atrophy (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify: perforated septum (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin and subcutaneous tissue disorders - Other, specify: Rash (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: Scrotum Rash (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: pressure ulcer (Skin and subcutaneous tissue disorders) | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Pheresis (Surgical and medical procedures) | 1
left brachial and axillary ulnar and radial thrombectomies (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT04493203/Prot_SAP_000.pdf